CLINICAL TRIAL: NCT06224452
Title: Is Ibrutinib-related Atrial Fibrillation Dose Dependent: Insights From the WHO Pharmacovigilance Database
Brief Title: Is Ibrutinib-related Atrial Fibrillation Dose Dependent
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco011624
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-01

CONDITIONS: Hematological Malignancy; Atrial Fibrillation
MeSH Terms: conditions — Hematologic Neoplasms; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: ibrutinib exposure — We will extract all atrial fibrillation cases involving adult patients associated with ibrutinib exposure with an available ibrutinib daily dose

SUMMARY:
Ibrutinib, an oral inhibitor of Bruton tyrosine kinase (BTK), has recently revolutionized the treatment of various chronic B-cell malignancies and particularly chronic lymphocytic leukemia (CLL). Atrial fibrillation (AF) has early emerged as a cardiovascular adverse effect (CVAE) of ibrutinib but underlying mechanisms of IRAF are not fully understood.

While a dose-reduction or an interruption of ibrutinib is mentioned in the summary of product characteristics of ibrutinib, any beneficial effect on IRAF management of such a management is unclear.

The main aim of this study is to determine if IRAF is a dose-dependent CVAE in chronic B-cell malignancies patients by studying the association between ibrutinib dose and IRAF reporting in Vigibase®, the World Health Organization (WHO) pharmacovigilance database.

DETAILED DESCRIPTION:
Ibrutinib, an oral inhibitor of Bruton tyrosine kinase (BTK), has recently revolutionized the treatment of various chronic B-cell malignancies and particularly chronic lymphocytic leukemia (CLL). Atrial fibrillation (AF) has early emerged as a cardiovascular adverse effect (CVAE) of ibrutinib. In phase 3 randomized clinical trials (RCT), ibrutinib exhibits a ≈4-fold increase-risk of AF compared with controls (pooled relative-risk (RR) 3.9; 95% confidence interval (CI): (2.0-7.5); p<0.0001). The annualized incidence rate of ibrutinib-related AF (IRAF) reporting in clinical trials is estimated to 4.9 (95% CI: 2.9-8.3) per 100 person-years. IRAF risk persists throughout ibrutinib exposition and seems to be cumulative with the extension of follow-up and cardiac monitoring.

Underlying mechanisms of IRAF are not fully understood. Ibrutinib potently inhibits multiple off-target kinases at therapeutic concentrations.

While a dose-reduction or an interruption of ibrutinib is mentioned in the summary of product characteristics of ibrutinib, any beneficial effect on IRAF management of such a management is unclear.

The main aim of this study is to determine if IRAF is a dose-dependent CVAE in chronic B-cell malignancies patients by studying the association between ibrutinib dose and IRAF reporting in Vigibase®, the World Health Organization (WHO) pharmacovigilance database.

ELIGIBILITY:
Inclusion Criteria:

* ibrutinib-related atrial fibrillation reports in Vigibase at the time of data extraction
* involving adult patients
* with an available ibrutinib daily dose

Exclusion Criteria:

* minors
* no ibrutinib dose available

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * ibrutinib-related atrial fibrillation reports in Vigibase at the time of data extraction
  * involving adult patients
  * with an available ibrutinib daily dose
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
to determine the influence of ibrutinib dosing on IRAF reporting. Results were expressed as 2-by2 comparisons against the lowest dosing regimen (140mg/day). | Cases reported in the World Health Organization (WHO) of individual safety case reports to 26th July 2023
  Disproportionality estimates will be perform using both univariate and multivariate analyses and a global p-value will measure the difference between dosing regimen

SECONDARY OUTCOMES:
Description of ibrutinib-related atrial fibrillation cases | Cases reported in the World Health Organization (WHO) of individual safety case reports to 26th July 2023
  Clinical caracteristics of ibrutinib-related atrial fibrillation cases (sex, age, time to onset, hematological malignacy, coreported drugs, coreported adverse events)
To determine the influence of ibrutinib dosing on IRAF reporting after exclusion of IRAF cases containing concurrent anticoagulant and/or antiarrhythmic drugs, assuming this approach could exclude reports with history of AF preceding IRAF reporting | Cases reported in the World Health Organization (WHO) of individual safety case reports to 26th July 2023
  Disproportionality estimates will be perform both univariate and multivariate analysesand a global p-value will measure the difference between dosing regimen
To determine the influence of ibrutinib dosing on IRAF reporting according to the underlying chronic B-cell malignancy indication. | Cases reported in the World Health Organization (WHO) of individual safety case reports to 26th July 2023
  Disproportionality estimates will be perform using both univariate and multivariate analyses and a global p-value will measure the difference between dosing regimen
To determine if the time to IRAF onset is dependent of the ibrutinib dosing regimen | Cases reported in the World Health Organization (WHO) of individual safety case reports to 26th July 2023
  We will use a linear regression to test if the association between ibrutinib-related atrial fibrillation reporting and time to onset is dependent of the dose regimen (the 140 mg/day ibrutinib dosing regimen will set as the reference)
Sensitivity analysis will also be performed regarding the influence of ibrutinib dosing on 2 dose-dependent ADRs (neutropenia and thrombocytopenia) reporting related to ibrutinib exposure | Cases reported in the World Health Organization (WHO) of individual safety case reports to 26th July 2023
  Disproportionality estimates will be perform using univariate analysis and a global p-value will measure the difference between dosing regimen

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Alexandre, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No
data are extracted from vigibase; data sharement is conditionned to the opinion of the Uppsala Monitoring Centre

REFERENCES:
- [Derived] Alexandre J, Font J, Angelique DS, Delapierre B, Damaj G, Plane AF, Legallois D, Milliez P, Dolladille C, Chretien B. Is ibrutinib-related atrial fibrillation dose dependent? Insights from an individual case level analysis of the World Health Organization pharmacovigilance database. Leukemia. 2024 Dec;38(12):2628-2635. doi: 10.1038/s41375-024-02413-5. Epub 2024 Sep 19. PMID 39300222